CLINICAL TRIAL: NCT04391634
Title: Cerebral Oxygenation and Circulatory Parameters During Pressure Controlled vs. Volume Targeted Mechanical Ventilation in the Extremely Preterm Infants With Respiratory Distress Syndrome
Brief Title: Cerebral and Circulatory Effects of Neonatal Volume Targeted Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 388/16
Record Dates: First submitted 2020-05-07; First posted 2020-05-18 (Actual); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Respiratory Distress Syndrome, Newborn; Respiratory Failure; Premature Birth
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Insufficiency; Premature Birth

STUDY DESIGN:
Intervention Model Description: prospective crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mechanical ventilation (Other): Preterm infants on mechanical ventilation
  Interventions: Other: volume guarantee; Other: pressure-controlled

INTERVENTIONS:
Other: volume guarantee — volume guarantee assist-control mechanical ventilation
Other: pressure-controlled — pressure-controlled assist-control mechanical ventilation

SUMMARY:
The aim of the study was to assess the effect of volume targeted vs. pressure-controlled mechanical ventilation (MV) on circulatory parameters and cerebral oxygenation in the extremely preterm infants.

DETAILED DESCRIPTION:
Prospective, cross-over trial enrolling neonates <28 weeks' gestation requiring MV. Patients were ventilated for 3 hours with pressure controlled assist-control (PC-AC) mode, followed by 3-hours of volume guarantee assist-control ventilation (VG-AC). Continuous monitoring was carried out using pulse oximetry (oxygen saturation - SpO2 and heart rate - HR), near-infrared spectroscopy (cerebral oxygenation - StO2) and electrical cardiometry (circulatory parameters).

ELIGIBILITY:
Inclusion Criteria:

* premature infants born <28 weeks of gestation
* respiratory failure in the course of respiratory distress syndrome requiring mechanical ventilation
* stable condition with pH (acidity of blood)> 7.2 and pCO2 (carbon dioxide partial pressure) <60 mmHg in the blood gas analysis
* no identified genetic syndromes and serious congenital malformations

Exclusion Criteria:

* lack of written consent of patients' parents

Ages: 24 Weeks to 27 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
StO2 | 6 hours
  Cerebral oxygenation measured using near-infrared spectroscopy [percent]
Stroke volume | 6 hours
  Stroke volume (SV) monitored with electrical cardiometry [ml]
Cardiac output | 6 hours
  Cardiac output (CO) monitored with electrical cardiometry [L/min]
Stroke index | 6 hours
  Stroke index (SI) monitored with electrical cardiometry [ml/m2]
Cardiac index | 6 hours
  Cardiac index (CI) monitored with electrical cardiometry [L/min/m2]
Stroke volume variation (SVV) | 6 hours
  Stroke volume variation (SVV) monitored with electrical cardiometry [percent]
Index of contractility | 6 hours
  Index of contractility (ICON) monitored with electrical cardiometry

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Szczapa, MD, PhD, Study Chair — Poznan University of Medical Sciences
Locations (1):
- Department of Neonatology at Poznań University of Medical Sciences, Poznan, Poland